CLINICAL TRIAL: NCT05719974
Title: Functional Outcomes of a Criterion-based Rehabilitation Protocol for Anterior Cruciate Ligament Reconstruction in Amateur Athlete: Randomized Controlled Trial
Brief Title: Functional Outcomes of a Criterion-based Rehabilitation Protocol for ACL Reconstruction in Amateur Athlete
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Deltau
Record Dates: First submitted 2023-01-28; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Knee Ligament Injury; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- criterion-based rehabilitation protocol (Experimental)
  Interventions: Other: rehabilitation protocol
- conventional physical therapy program (Active Comparator)
  Interventions: Other: rehabilitation protocol

INTERVENTIONS:
Other: rehabilitation protocol — Current conventional protocols were based mainly on biological tissue healing time frames. These protocols emphasize pain reduction, full passive knee extension, quadriceps strength training, immediate motion, immediate par¬tial weight bearing (only if there is a correct gait pattern without any complications), and functional exercises The criterion-based rehabilitation protocol is relatively new. It was developed and recommended in 2016 by the Royal Dutch Society for Physical Therapy (KNGF), aiming to assure a more patient-tailored rehabilitation and to maximize the speed of a patient's progress. It's a three phases protocol with a criterion-based progression.

SUMMARY:
Although current rehabilitation protocols following anterior cruciate ligament reconstruction (ACLR) are based on the graft remodeling process, there is uncertainty about its time schedule. Moreover, there are individual differences in neuromotor learning and flexibility after ACLR. This study was conducted to investigate the effect of a criterion-based rehabilitation protocol on pain intensity, effusion, and knee function in amateur athletes following ACLR.

Although current rehabilitation protocols following anterior cruciate ligament reconstruction (ACLR) are based on the graft remodeling process, there is uncertainty about its time schedule. Moreover, there are individual differences in neuromotor learning and flexibility after ACLR. This study was conducted to investigate the effect of a criterion-based rehabilitation protocol on pain intensity, effusion, and knee function in amateur athletes following ACLR.

ELIGIBILITY:
Inclusion Criteria:

* Amateur male athletes who underwent ACLR surgery with an autologous hamstring (HS) graft.
* Ranging in age from 18 to 35 years.
* Underwent a pre-operative rehabilitation program with minimal knee effusion, full Extension, good patellofemoral mobility
* Ability to actively control the quadriceps.

Exclusion Criteria:

* ACLR with any graft other than a hamstring graft
* ACL revision surgery
* associated medial or lateral ligamentous injuries
* previous meniscectomy or meniscal repair
* simultaneous meniscectomy or meniscus repair with the ACLR
* cartilage damage.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 months
  It is a 100-mm horizontal line anchored by word descriptors at each end by "no pain" on the left and "worst imaginable pain" on the right

SECONDARY OUTCOMES:
limb symmetry index of hop test battery | 6 months
  The mean score of the results of each item of hop test battery of the injured limb was divided by the corresponding mean score of the uninjured limb and the result was multiplied by 100. Hop test battery consists of the following: (1) vertical jump, (2) hop for distance, (3) drop jump followed by a double hop for distance, (4) square hop and (5) side hop.
Knee Injury and Osteoarthritis Outcome Score | 6 months
  it is a 42-item self-questionnaire with five subscales. A five-point scale ranging from 0 (no problem) to 4 (extreme problems) was used to score each item and the scores of each subscale were individually transformed into a 0-100 scale (0 = extreme knee problems, 100 = no knee problem)
knee effusion grading scale | 6 months
  It"s a reliable and valid method which Based on a stroke test, where effusion of the knee joint is quantified using a 5-point scale. A 0 grade means no wave is produced with the downward stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university, Gamasa, Eldakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No